CLINICAL TRIAL: NCT04138953
Title: Characterizing Cortical Contributions to Motor Sequence Learning
Brief Title: Cortical Contributions to Motor Sequence Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Michael R Borich, Assitant professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00115009
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Brain Injuries
Keywords: Electrophysiology; Magnetic Resonance imaging (MRI); Neuroanatomy; Neuroscience
MeSH Terms: conditions — Brain Injuries | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- TMS over premotor cortex (PMC) (Experimental): Noninvasive brain stimulation in the premotor cortex
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- TMS over primary motor cortex (M1) (Experimental): Noninvasive brain stimulation in the motor cortex
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Sham TMS (Sham Comparator): Sham brain stimulation
  Interventions: Other: Sham TMS

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Transcranial magnetic stimulation, also known as repetitive transcranial magnetic stimulation, is a noninvasive form of brain stimulation in which a changing magnetic field is used to cause electric current at a specific area of the brain through electromagnetic induction.
  It will be used to create a 'virtual lesion,' disrupting neural activity in a specific brain region to identify whether it is causally involved in a specific behavioral process.
  Other Names: TMS
  Arms: TMS over premotor cortex (PMC); TMS over primary motor cortex (M1)
Other: Sham TMS — Sham Transcranial Magnetic Stimulation (TMS)
  Arms: Sham TMS

SUMMARY:
The long-term objective initiated with this study is to determine which brain areas functionally contribute to learning a motor skill. The primary hypothesis of this trial is that premotor cortex (PMC) is necessary to learn a new motor skill. Participants may undergo a MRI scan to acquire a structural image of their brain to target noninvasive stimulation, using transcranial magnetic stimulation (TMS) to one of two brain areas: PMC or primary motor cortex (M1). A third group of individuals will undergo a placebo stimulation protocol. For all three groups, stimulation will be used to create a transient 'virtual lesion' during motor skill training. Temporarily disrupting the normal activity of these brain regions during training will allow us to determine which regions are causally involved in learning a new motor skill. The primary outcome measure will be the change in skill after training in each group.

DETAILED DESCRIPTION:
Recent findings in humans suggest that motor sequences are represented in the premotor cortex once learned. Studies in animal models have also shown that the premotor cortical areas encode sequence-specific information. However, it is currently unknown if premotor cortical areas are involved in the acquisition or consolidation of sequences in humans. In this project, the investigators will evaluate the functional contributions of human premotor cortex to sequence learning. The primary overarching research objective is to determine the brain regions causally involved in motor skill acquisition and consolidation. The main hypothesis is that disrupting premotor cortex activity during motor sequence learning will reduce the acquisition and consolidation of the skill. Transcranial magnetic stimulation (TMS) will be used to temporarily disrupt activity of premotor cortex or primary motor cortex, and skill learning will be assessed in both groups. A sham stimulation group, where participants will feel the coil on their head and hear the click of the TMS pulses but not actually receive stimulation to the brain, will be used as a control. Participants will be randomly assigned to be in the premotor cortex, primary motor cortex, or sham stimulation group. Participants may be asked to undergo a Magnetic Resonance Imaging (MRI) scan at Wesley Woods prior to TMS testing, which will occur at the Emory Rehabilitation Hospital. The MRI scan would be used to help target TMS to the intended brain area. Participants will be recruited using flyers around the local community. Consent forms will be provided with ample time for the participant to read it over and ask any questions that may arise. Participants will be compensated for their time. The proposed work will be the first to evaluate the causal role of premotor cortex in motor sequence learning in humans. Findings from this project are expected to inform the design and application of therapeutic interventions that improve motor functioning and learning in clinical populations.

ELIGIBILITY:
Inclusion Criteria:

* No history of movement impairment or neurodegenerative disease
* Right handedness
* No contraindication to transcranial magnetic stimulation (TMS) or magnetic resonance imaging (MRI).

Exclusion Criteria:

* Participants that are outside the age range of 18-85
* Have a history of head trauma or neurodegenerative disorder
* Report contraindications to TMS.
* Participants over age 65 will be asked to complete the Montreal Cognitive Assessment, and participants with a score of 25 or lower (out of the "normal" range) will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Borich, DPT, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Wesley Woods, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Neurophysiology and motor performance outcome measures will be shared
Supporting Information: Study Protocol, SAP
Time Frame: . Data will be available after publication of primary study results (estimated 12 months after study completion - no end date specified)
Access Criteria: Data will be shared through secure file transfer to researchers requesting access to data collected as part of this study

RESULTS

PARTICIPANT FLOW:
Groups:
- TMS Over Primary Motor Cortex (M1): Noninvasive brain stimulation in the motor cortex
  Transcranial Magnetic Stimulation (TMS): Transcranial magnetic stimulation, also known as repetitive transcranial magnetic stimulation, is a noninvasive form of brain stimulation in which a changing magnetic field is used to cause electric current at a specific area of the brain through electromagnetic induction.
  It will be used to create a 'virtual lesion,' disrupting neural activity in a specific brain region to identify whether it is causally involved in a specific behavioral process.
- TMS Over Premotor Cortex (PMC): Noninvasive brain stimulation in the premotor cortex
  Transcranial Magnetic Stimulation (TMS): Transcranial magnetic stimulation, also known as repetitive transcranial magnetic stimulation, is a noninvasive form of brain stimulation in which a changing magnetic field is used to cause electric current at a specific area of the brain through electromagnetic induction.
  It will be used to create a 'virtual lesion,' disrupting neural activity in a specific brain region to identify whether it is causally involved in a specific behavioral process.
Period: Overall Study
Arm/Group | Sham TMS | TMS Over Primary Motor Cortex (M1) | TMS Over Premotor Cortex (PMC)
Started | 20 | 20 | 24
Completed | 20 | 20 | 24
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham TMS | TMS Over Primary Motor Cortex (M1) | TMS Over Premotor Cortex (PMC) | Total
Number analyzed (Participants) | 20 | 20 | 24 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 24 | 64
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 16 | 42
  Male | 8 | 6 | 8 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Pacific Islander | 5 | 1 | 4 | 10
  Black or African American | 0 | 0 | 2 | 2
  Hispanic or Latino | 1 | 3 | 1 | 5
  White | 11 | 13 | 15 | 39
  Multi racial | 1 | 2 | 1 | 4
  Unknown | 2 | 1 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 24 | 64

OUTCOME MEASURES:

1. Primary Outcome: Serial Reaction Time Task (SRTT) Performance
Description: The SRTT involves pressing a key that corresponds to a target square presented on a monitor. Sequenced skill (SS) is calculated by subtracting the response time of sequenced key presses from random key presses within and across a test block. An increase in SS value indicates an increase in sequenced skill and is a preferable result.
Time Frame: Pre-test (baseline), Post-test (training usually lasts for 3 hours), Retention Test (30 mins following training)
Population: The population in this analysis includes participants who completed the indicated study visit and had usable data. Five participants in the PMC group are not included due to technical issues; for 2 participants the stimulation target could not be confirmed during data analysis and 3 participants had different timing values than other members of their cohort. Of participants with usable pre- and post- test data, 11 from the M1 group and 12 from the PMC group completed the retention test.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Sham TMS | TMS Over Primary Motor Cortex (M1) | TMS Over Premotor Cortex (PMC)
Number analyzed (Participants) | 20 | 20 | 19
milliseconds (ms)
  SS Pre-test | 31 (38) | 35 (19) | 38 (24)
  SS Post-test | 24 (21) | 30 (22) | 17 (23)
  SS Retention Testing: number analyzed (Participants) | 20 | 11 | 12
  SS Retention Testing | 31 (25) | 40 (23) | 29 (11)

2. Secondary Outcome: Cortical Excitability Measured by Motor Evoked Potentials (MEPs)
Description: Evaluate the effect of sequence learning on motor cortical excitability. Cortical excitability will be indexed by peak-to-peak amplitudes of transcranial magnetic stimulation (TMS)-evoked electromyographic responses in the hand contralateral to the motor cortex targeted by TMS quantified before and after training. An increase in MEPs indicates neural plasticity due to increases in skill.
Time Frame: Pre-test (baseline), Post-test (training usually lasts for 3 hours)
Population: The population in this analysis includes participants who completed the indicated study visit and had usable data. Five participants in the premotor cortex (PMC) group are not included due to technical issues; for two participants the stimulation target could not be confirmed during data analysis and three participants had different timing values than other members of their cohort.
Measure: Mean (Standard Deviation); unit: millivolts (mV)
Arm/Group | Sham TMS | TMS Over Primary Motor Cortex (M1) | TMS Over Premotor Cortex (PMC)
Number analyzed (Participants) | 20 | 20 | 19
millivolts (mV)
  MEP Amplitude Pre-test | 1.03 (0.97) | 1.29 (1.22) | 0.45 (0.37)
  MEP Amplitude Post-test | 1.15 (1.03) | 1.37 (1.24) | 0.51 (0.53)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the entire duration of participation, from the time of informed consent through completing the retention testing, up to 28 hours.
Arm/Group | Sham TMS | TMS Over Primary Motor Cortex (M1) | TMS Over Premotor Cortex (PMC)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/24
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT04138953/Prot_SAP_000.pdf